CLINICAL TRIAL: NCT07057180
Title: The Impact of Intensive Care Nurses' Caring Behaviors on the Quality of Nursing Care
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Saadet Can Çiçek, Associate Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-SBF-NSS-25
Record Dates: First submitted 2025-06-12; First posted 2025-07-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Perception of Caring Behaviors; Quality of Nursing Care
Keywords: Perception of Caring Behaviors; Quality of Nursing Care; Intensive Care; Intensive Care Nurse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples Without DNA — 'Nursing Comprehensive Care Observation Form' and 'Nurses' care-related behaviors and perceptions as evaluated through self-assessment'
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive Care Unit (ICU) Nurses: Nurses who have been working in intensive care units for at least 3 months with a registered nurse title,
  Nurses who have provided verbal and written informed consent to participate in the study,
  Nurses who are rotationally responsible for patient populations whose care quality is evaluated during 24-hour shifts.
  Interventions: Behavioral: This involves nurses' self-assessment of their caregiving behaviors and perceptions
- Patients admitted to the Intensive Care Unit (ICU): Patients aged 18 years and older,
  Patients whose legal representatives have provided verbal and written informed consent for participation,
  Patients with a Foley catheter in place for a minimum of 14 days, as urine bag replacement is evaluated after this period,
  Patients who are intubated, mechanically ventilated, possess invasive catheters for nutrition and monitoring, and are fully dependent on nursing care.
  Interventions: Other: Observation by the Researcher and Self-evaluations by nurses

INTERVENTIONS:
Other: Observation by the Researcher and Self-evaluations by nurses — Observation by the Researcher
  Groups: Patients admitted to the Intensive Care Unit (ICU)
Behavioral: This involves nurses' self-assessment of their caregiving behaviors and perceptions — This refers to the clinical observation performed by the nurse researcher
  Groups: Intensive Care Unit (ICU) Nurses

SUMMARY:
Brief Summary The purpose of this observational study is to find out whether the caring behaviors of intensive care nurses affect the quality of nursing care for adult patients in the Intensive Care Unit (ICU) at Bolu Izzet Baysal State Hospital.

The study aims to answer the following questions:

Do nurses' caring behaviors influence the quality of care that patients receive?

Are nurses' personal and professional characteristics related to their caring behaviors and the quality of care?

In this study:

Nurses will complete questionnaires about their caring behaviors and personal information.

The researcher will observe patients and assess the quality of care they receive.

The study will be conducted between June 1, 2025, and June 1, 2026. The results are expected to support training programs and improvement efforts to enhance nursing care quality in ICUs.

DETAILED DESCRIPTION:
This observational study investigates whether the caring behaviors of intensive care nurses influence the quality of nursing care for adult patients in the intensive care unit (ICU) at Bolu Izzet Baysal State Hospital.

Nurses play a critical role in providing continuous, high-quality care to critically ill patients. Research suggests that nurses' behaviors and communication can significantly affect patient care experiences and outcomes.

Based on clinical observations, variations in the perceived quality of care have been noticed, especially during shift changes in the ICU. This study aims to assess both how nurses perceive their caring behaviors and how the quality of care is observed by the researcher.

Findings from the study are expected to help identify areas for improvement and inform potential training programs to enhance care quality, teamwork, and communication within ICU settings.

ELIGIBILITY:
Inclusion Criteria for Nurses:

Registered nurses who have been working in intensive care units for at least 3 months,

Nurses who have provided both verbal and written informed consent to participate in the study,

Nurses who are rotationally responsible for patient populations whose nursing care quality is assessed during 24-hour shifts.

Inclusion Criteria for Patients:

Patients aged 18 years or older,

Patients whose legal guardians have provided verbal and written informed consent to participate in the study,

Patients with a Foley catheter in place for a minimum of 14 days, as this duration is required to evaluate urinary catheter management quality,

Patients who are intubated, mechanically ventilated, equipped with invasive catheters for nutrition and monitoring, and are fully dependent on nursing care.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and above, admitted to the intensive care unit and meeting the study's inclusion criteria and Intensive Care Unit (ICU) Nurses
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Total score of the Caring Behaviors Inventory-24 (CBI-24) completed by ICU nurses | Each nurse will complete the questionnaire once during the study period
  The CBI-24 consists of 24 items rated on a 6-point Likert scale (1 = Never, 6 = Always). Higher total scores indicate higher levels of self-perceived caring behaviors by ICU nurses. Due to the rotational shift system, all ICU nurses contribute to the care of multiple patients over time. Therefore, each nurse will complete the questionnaire only once during the study period to capture their overall perception of caring behaviors.

SECONDARY OUTCOMES:
Total score of the "Quality of Nursing Care in Intensive Care Units Scale" assessed by the researcher through bedside observation | Data collected during each patient's stay in the ICU
  The scale includes 50 items rated on a 3-point Likert scale (0 = Not satisfactory, 2 = Highly satisfactory). Total scores range from 0 to 100. Higher scores indicate better nursing care quality as assessed by the researcher.

OTHER OUTCOMES:
Comparison of ICU nurses' self-perceived caring behaviors (CBI-24 total score) and nursing care quality (Quality Scale total score) | Analyzed after completion of data collection
  The relationship between ICU nurses' self-perceived caring behaviors (CBI-24 total scores) and nursing care quality scores observed by the researcher will be evaluated using linear regression analysis. The goal is to determine whether higher caring behaviors are associated with higher nursing care quality.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Republic of Turkey, Ministry of Health, Bolu Izzet Baysal State Hospital, Merkez, Bolu
  - Bolu Abant Izzet Baysal Unıversıtesı, Bolu

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to ethical considerations.